CLINICAL TRIAL: NCT02031640
Title: A Randomized, Double-Blind, Double-Dummy, Placebo Controlled, Parallel-Group, 12-Week Clinical Study to Assess the Efficacy and Safety of 320 or 640 mcg/Day of Beclomethasone Dipropionate Delivered Via Breath-Actuated Inhaler (BAI) or Metered-Dose Inhaler (MDI) in Adolescent and Adult Patients 12 Years of Age and Older With Persistent Asthma
Brief Title: A Safety and Efficacy Study of Beclomethasone Dipropionate Delivered Via Breath-Actuated Inhaler (BAI) or Metered-Dose Inhaler (MDI) in Participants >=12 Years Old With Persistent Asthma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BDB-AS-301; 2013-003397-27 (EudraCT Number)
Record Dates: First submitted 2014-01-07; First posted 2014-01-09 (Estimated); Results first posted 2018-01-05 (Actual); Last update posted 2021-11-09 (Actual); Status verified 2021-11

CONDITIONS: Asthma
Keywords: asthma; breath-actuated inhaler; metered-dose inhaler
MeSH Terms: conditions — Asthma | interventions — Beclomethasone; Albuterol; Bronchodilator Agents

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- BDP 320 mcg BAI (Experimental): Beclomethasone dipropionate (BDP) via breath-actuated inhaler (BAI) twice daily.
  Interventions: Drug: Beclomethasone dipropionate; Drug: Placebo; Drug: Albuterol/salbutamol
- BDP 640 mcg BAI (Experimental): Beclomethasone dipropionate (BDP) via breath-actuated inhaler (BAI) twice daily.
  Interventions: Drug: Beclomethasone dipropionate; Drug: Placebo; Drug: Albuterol/salbutamol
- BDP 320 mcg MDI (Active Comparator): Beclomethasone dipropionate (BDP) via metered dose inhaler (MDI) twice daily.
  Interventions: Drug: Beclomethasone dipropionate; Drug: Placebo; Drug: Albuterol/salbutamol
- BDP 640 mcg MDI (Active Comparator): Beclomethasone dipropionate (BDP) via metered dose inhaler (MDI) twice daily.
  Interventions: Drug: Beclomethasone dipropionate; Drug: Placebo; Drug: Albuterol/salbutamol
- Placebo BAI and MDI (Placebo Comparator): Placebo breath-actuated inhaler (BAI), twice daily. Plus placebo metered dose inhaler (MDI), twice daily.
  Interventions: Drug: Placebo; Drug: Albuterol/salbutamol

INTERVENTIONS:
Drug: Beclomethasone dipropionate
  Other Names: BDP
  Arms: BDP 320 mcg BAI; BDP 320 mcg MDI; BDP 640 mcg BAI; BDP 640 mcg MDI
Drug: Placebo
Drug: Albuterol/salbutamol — Rescue medication (albuterol/salbutamol hydrofluoroalkane (HFA) MDI [90 mcg ex-actuator] or equivalent) for use on an as-needed basis for the immediate relief of asthma symptoms throughout the treatment period.
  Other Names: bronchodilators

SUMMARY:
This is a Phase 3, randomized, placebo-controlled, double-blind,double-dummy, parallel-group, 12-week study in male and female patients, 12 years of age and older, with persistent asthma.

ELIGIBILITY:
Inclusion Criteria:

* Severity of disease: The patient has persistent asthma, with a forced expiratory volume in 1 second (FEV1) 40%-85% of the value predicted for age, height, sex, and race as per the National Health and Nutrition Examination Survey (NHANES III) (Hankinson et al 1999) reference values at screening visit.
* Current asthma therapy: The patient must be on a stable dose of an inhaled corticosteroid (ICS) of at least 440 mcg/day of fluticasone propionate or equivalent for a minimum of 4 weeks before screening visit, or any inhaled corticosteroid/long-acting beta2-agonist (ICS/LABA) combination for a minimum of 4 weeks before the prescreening visit.
* Reversibility of disease: The patient has demonstrated at least 12% reversibility of FEV1 and at least 200 mL increase from baseline FEV1 (patients age 18 and older) within 30 minutes after 2-4 inhalations of albuterol/salbutamol hydrofluoroalkane (HFA) MDI (90 mcg ex-actuator) or equivalent at the screening visit
* If female, the patient is currently not pregnant, breast feeding, or attempting to become pregnant. If of childbearing potential, has a negative serum pregnancy test and is willing to commit to using a consistent and acceptable method of birth control.
* Other criteria apply, please contact the investigator for more information

Exclusion Criteria:

* The patient has a history of life-threatening asthma, defined for this protocol as an asthma episode that required intubation and/or was associated with hypercapnea, respiratory arrest, or hypoxic seizures.
* The patient is pregnant or lactating, or plans to become pregnant during the study period or for 30 days after the patient's last study-related visit (for eligible patients only, if applicable). Eligible female patients unwilling to employ appropriate contraceptive measures to ensure that pregnancy will not occur during the study will be excluded. Any patient becoming pregnant during the study will be withdrawn from the study.
* The patient has a known hypersensitivity to any corticosteroid or any of the excipients in the study drug or rescue medication formulation.
* The patient currently smokes or has a smoking history of 10 pack-years or more (a pack-year is defined as smoking 1 pack of cigarettes/day for 1 year).
* The patient has had an asthma exacerbation requiring oral corticosteroids within 30 days before the screening visit, or has had any hospitalization for asthma within 2 months before the screening visit.
* The patient has historical or current evidence of a clinically significant disease. Significant disease is defined as any disease that in the medical judgment of the investigator would put the safety of the patient at risk through participation or that could affect the efficacy or safety analysis if the disease/condition worsened during the study.
* Other criteria apply, please contact the investigator for more information

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1113 (Actual)
Dates: Start 2013-12; Primary Completion 2014-11 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Teva Medical Expert, MD, Study Director — Teva Branded Pharmaceutical Products R&D, Inc.
Locations (131):
- United States (94):
  - Teva Investigational Site 10851, Costa Mesa, California
  - Teva Investigational Site 10849, Huntington Beach, California
  - Teva Investigational Site 10872, Huntington Beach, California
  - Teva Investigational Site 10833, Long Beach, California
  - Teva Investigational Site 10861, Los Angeles, California
  - Teva Investigational Site 10798, Mission Viejo, California
  - Teva Investigational Site 10806, Orange, California
  - Teva Investigational Site 10828, Orange, California
  - Teva Investigational Site 10860, Paramount, California
  - Teva Investigational Site 10813, Rancho Mirage, California
  - Teva Investigational Site 10843, Riverside, California
  - Teva Investigational Site 10857, Rolling Hills Estates, California
  - Teva Investigational Site 10847, San Diego, California
  - Teva Investigational Site 10871, San Diego, California
  - Teva Investigational Site 10876, San Jose, California
  - Teva Investigational Site 12270, Walnut Creek, California
  - Teva Investigational Site 12266, Centennial, Colorado
  - Teva Investigational Site 10838, Colorado Springs, Colorado
  - Teva Investigational Site 10844, Denver, Colorado
  - Teva Investigational Site 10799, Wheat Ridge, Colorado
  - Teva Investigational Site 10826, Aventura, Florida
  - Teva Investigational Site 10877, Clearwater, Florida
  - Teva Investigational Site 10816, Edgewater, Florida
  - Teva Investigational Site 12268, Melbourne, Florida
  - Teva Investigational Site 10807, Miami, Florida
  - Teva Investigational Site 10840, Miami, Florida
  - Teva Investigational Site 12269, Miami, Florida
  - Teva Investigational Site 10875, Sarasota, Florida
  - Teva Investigational Site 10855, Tallahassee, Florida
  - Teva Investigational Site 10864, Tampa, Florida
  - Teva Investigational Site 10858, Albany, Georgia
  - Teva Investigational Site 10862, Lawrenceville, Georgia
  - Teva Investigational Site 10848, Savannah, Georgia
  - Teva Investigational Site 10829, River Forest, Illinois
  - Teva Investigational Site 10809, Indianapolis, Indiana
  - Teva Investigational Site 10795, Iowa City, Iowa
  - Teva Investigational Site 10870, Owensboro, Kentucky
  - Teva Investigational Site 10832, Baltimore, Maryland
  - Teva Investigational Site 10850, Bethesda, Maryland
  - Teva Investigational Site 10873, Wheaton, Maryland
  - Teva Investigational Site 12272, White Marsh, Maryland
  - Teva Investigational Site 10834, North Dartmouth, Massachusetts
  - Teva Investigational Site 10815, Minneapolis, Minnesota
  - Teva Investigational Site 10821, Minneapolis, Minnesota
  - Teva Investigational Site 10869, Columbia, Missouri
  - Teva Investigational Site 10868, Rolla, Missouri
  - Teva Investigational Site 10867, St Louis, Missouri
  - Teva Investigational Site 12271, St Louis, Missouri
  - Teva Investigational Site 10827, Warrensburg, Missouri
  - Teva Investigational Site 12261, Missoula, Montana
  - Teva Investigational Site 10794, Bellevue, Nebraska
  - Teva Investigational Site 10814, Bellevue, Nebraska
  - Teva Investigational Site 10846, Brick, New Jersey
  - Teva Investigational Site 10817, Marlton, New Jersey
  - Teva Investigational Site 10856, Ocean City, New Jersey
  - Teva Investigational Site 10845, Skillman, New Jersey
  - Teva Investigational Site 10801, Rochester, New York
  - Teva Investigational Site 10842, Canton, Ohio
  - Teva Investigational Site 10792, Cincinnati, Ohio
  - Teva Investigational Site 10811, Cincinnati, Ohio
  - Teva Investigational Site 10874, Sylvania, Ohio
  - Teva Investigational Site 12265, Toledo, Ohio
  - Teva Investigational Site 10800, Oklahoma City, Oklahoma
  - Teva Investigational Site 10853, Oklahoma City, Oklahoma
  - Teva Investigational Site 10865, Oklahoma City, Oklahoma
  - Teva Investigational Site 12796, Oklahoma City, Oklahoma
  - Teva Investigational Site 10818, Tulsa, Oklahoma
  - Teva Investigational Site 10822, Eugene, Oregon
  - Teva Investigational Site 10791, Lake Oswego, Oregon
  - Teva Investigational Site 10824, Medford, Oregon
  - Teva Investigational Site 10835, Portland, Oregon
  - Teva Investigational Site 10859, Philadelphia, Pennsylvania
  - Teva Investigational Site 12795, Warwick, Rhode Island
  - Teva Investigational Site 10837, North Charleston, South Carolina
  - Teva Investigational Site 12262, Orangeburg, South Carolina
  - Teva Investigational Site 10803, Knoxville, Tennessee
  - Teva Investigational Site 10820, Austin, Texas
  - Teva Investigational Site 10808, Boerne, Texas
  - Teva Investigational Site 10830, Dallas, Texas
  - Teva Investigational Site 10831, El Paso, Texas
  - Teva Investigational Site 10878, Live Oak, Texas
  - Teva Investigational Site 10810, Plano, Texas
  - Teva Investigational Site 10797, San Antonio, Texas
  - Teva Investigational Site 10812, San Antonio, Texas
  - Teva Investigational Site 10793, Sugar Land, Texas
  - Teva Investigational Site 10790, Waco, Texas
  - Teva Investigational Site 10823, South Burlington, Vermont
  - Teva Investigational Site 10796, Richmond, Virginia
  - Teva Investigational Site 10854, Richmond, Virginia
  - Teva Investigational Site 10805, Bellingham, Washington
  - Teva Investigational Site 10866, Seattle, Washington
  - Teva Investigational Site 12264, Tacoma, Washington
  - Teva Investigational Site 10863, Greenfield, Wisconsin
  - Teva Investigational Site 10836, Madison, Wisconsin
- Germany (11):
  - Teva Investigational Site 32326, Berlin
  - Teva Investigational Site 32332, Berlin
  - Teva Investigational Site 32334, Berlin
  - Teva Investigational Site 32331, Frankfurt
  - Teva Investigational Site 32335, Gelnhausen
  - Teva Investigational Site 32329, Leipzig
  - Teva Investigational Site 32330, Magdeburg
  - Teva Investigational Site 32333, Mainz
  - Teva Investigational Site 32327, Munich
  - Teva Investigational Site 32328, München
  - Teva Investigational Site 32325, Rüdersdorf
- Hungary (10):
  - Teva Investigational Site 51081, Budapest
  - Teva Investigational Site 51083, Debrecen
  - Teva Investigational Site 51084, Debrecen
  - Teva Investigational Site 51080, Érd
  - Teva Investigational Site 51108, Győr
  - Teva Investigational Site 51079, Kapuvár
  - Teva Investigational Site 51109, Komárom
  - Teva Investigational Site 51086, Nyíregyháza
  - Teva Investigational Site 51078, Siófok
  - Teva Investigational Site 51087, Szombathely
- Poland (16):
  - Teva Investigational Site 53121, Bialystok
  - Teva Investigational Site 53129, Bialystok
  - Teva Investigational Site 53130, Bialystok
  - Teva Investigational Site 53154, Gdansk
  - Teva Investigational Site 53155, Katowice
  - Teva Investigational Site 53124, Krakow
  - Teva Investigational Site 53125, Lodz
  - Teva Investigational Site 53132, Lodz
  - Teva Investigational Site 53126, Lubin
  - Teva Investigational Site 53157, Lublin
  - Teva Investigational Site 53122, Ostrów Wielkopolski
  - Teva Investigational Site 53156, Poznan
  - Teva Investigational Site 53123, Strzelce Opolskie
  - Teva Investigational Site 53127, Tarnów
  - Teva Investigational Site 53131, Warsaw
  - Teva Investigational Site 53128, Wroclaw

REFERENCES:
- [Derived] Amar NJ, Moss MH, Kerwin EM, Li J, Small CJ. Safety and efficacy of beclomethasone dipropionate delivered by breath-actuated or metered-dose inhaler for persistent asthma. Allergy Asthma Proc. 2016 Sep;37(5):359-69. doi: 10.2500/aap.2016.37.3983. Epub 2016 Aug 9. PMID 27510595

RESULTS

PARTICIPANT FLOW:
Recruitment Details: For this study, 125 sites were activated, 115 sites screened at least 1 patient (91 centers in the United States, 10 centers in Germany, 10 centers in Hungary, and 4 centers in Poland), and 97 sites randomized at least 1 patient.
Pre-assignment Details: There were two periods prior to treatment assignment: a screening period and a run-in period.
Groups:
- Consented Patients - Standard ICS and Placebo: Consented patients were placed on a standard inhaled corticosteroids (ICS) of fluticasone propionate through the Screening and Run-In Periods. The assigned total daily dose was 440 mcg/day or 880 mcg/day dependent upon prestudy asthma treatment.
  In addition to standard ICS, participants were provided with single-blind placebo BAI and single-blind placebo MDI device for twice-daily use during the Run-In period.
  Rescue medication (albuterol/salbutamol hydrofluoroalkane (HFA) metered dose inhaler (MDI) [90 mcg ex-actuator] or equivalent) for use on an as-needed basis for the immediate relief of asthma symptoms
- Placebo BAI and MDI: Placebo breath-actuated inhaler (BAI), twice daily. Plus placebo metered dose inhaler (MDI), twice daily.
  Rescue medication (albuterol/salbutamol hydrofluoroalkane (HFA) MDI [90 mcg ex-actuator] or equivalent) for use on an as-needed basis for the immediate relief of asthma symptoms.
- BDP 320 mcg BAI; BDP 640 mcg BAI: Beclomethasone dipropionate (BDP) via breath-actuated inhaler (BAI) twice daily.
  Placebo MDI for blinding.
  Rescue medication (albuterol/salbutamol hydrofluoroalkane (HFA) MDI [90 mcg ex-actuator] or equivalent) for use on an as-needed basis for the immediate relief of asthma symptoms.
- BDP 320 mcg MDI; BDP 640 mcg MDI: Beclomethasone dipropionate (BDP) via metered dose inhaler (MDI) twice daily.
  Placebo BAI for blinding.
  Rescue medication (albuterol/salbutamol hydrofluoroalkane (HFA) MDI [90 mcg ex-actuator] or equivalent) for use on an as-needed basis for the immediate relief of asthma symptoms.
Period: Screening Period
Arm/Group | Consented Patients - Standard ICS and Placebo | Placebo BAI and MDI | BDP 320 mcg BAI | BDP 640 mcg BAI | BDP 320 mcg MDI | BDP 640 mcg MDI
Started | 1113 (Consented) | 0 | 0 | 0 | 0 | 0
Completed | 701 | 0 | 0 | 0 | 0 | 0
Not Completed | 412 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 29 | 0 | 0 | 0 | 0 | 0
Not completed — Inclusion criteria not met | 312 | 0 | 0 | 0 | 0 | 0
Not completed — Exclusion criteria met | 30 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 14 | 0 | 0 | 0 | 0 | 0
Not completed — Enrollment closed | 26 | 0 | 0 | 0 | 0 | 0
Period: Run-In Period
Arm/Group | Consented Patients - Standard ICS and Placebo | Placebo BAI and MDI | BDP 320 mcg BAI | BDP 640 mcg BAI | BDP 320 mcg MDI | BDP 640 mcg MDI
Started | 701 | 0 | 0 | 0 | 0 | 0
Completed | 532 | 0 | 0 | 0 | 0 | 0
Not Completed | 169 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 4 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 17 | 0 | 0 | 0 | 0 | 0
Not completed — Inclusion criteria not met | 38 | 0 | 0 | 0 | 0 | 0
Not completed — Exclusion criteria met | 8 | 0 | 0 | 0 | 0 | 0
Not completed — Randomization criteria not met | 85 | 0 | 0 | 0 | 0 | 0
Not completed — Various administrative reasons | 17 | 0 | 0 | 0 | 0 | 0
Period: Double-blind Treatment Period
Arm/Group | Consented Patients - Standard ICS and Placebo | Placebo BAI and MDI | BDP 320 mcg BAI | BDP 640 mcg BAI | BDP 320 mcg MDI | BDP 640 mcg MDI
Started | 0 | 106 | 106 | 106 | 107 | 107
Full Analysis Set (Randomized patients with at least 1 dose of drug and 1 postbaseline trough am FEV1) | 0 | 106 | 104 | 106 | 106 | 107
Completed | 0 | 84 | 100 | 99 | 96 | 104
Not Completed | 0 | 22 | 6 | 7 | 11 | 3
Not completed — Protocol deviation | 0 | 2 | 0 | 1 | 3 | 1
Not completed — Lack of Efficacy | 0 | 14 | 3 | 2 | 5 | 1
Not completed — Non-compliance | 0 | 1 | 0 | 1 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 2 | 3 | 1 | 1 | 1
Not completed — Lost to Follow-up | 0 | 3 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Patients administered 4 inhalations from each of the 2 devices twice daily as per the double dummy study design: 1 treatment device or placebo and 1 placebo device for a total of 8 inhalations each time.
Groups:
- Placebo BAI and MDI: Placebo breath-actuated inhaler (BAI), twice daily. Plus placebo metered dose inhaler (MDI), twice daily.
  Rescue medication (albuterol/salbutamol hydrofluoroalkane (HFA) MDI [90 mcg ex-actuator] or equivalent) for use on an as-needed basis for the immediate relief of asthma symptoms throughout the treatment period.
- BDP 320 mcg BAI: Beclomethasone dipropionate (BDP) via breath-actuated inhaler (BAI) twice daily.
  Placebo MDI for blinding.
  Rescue medication (albuterol/salbutamol hydrofluoroalkane (HFA) MDI [90 mcg ex-actuator] or equivalent) for use on an as-needed basis for the immediate relief of asthma symptoms throughout the treatment period.
- BDP 640 mcg BAI: Beclomethasone dipropionate (BDP) via breath-actuated inhaler (BAI) twice daily.
  Placebo MDI for blinding.
  Albuterol/salbutamol: Rescue medication (albuterol/salbutamol hydrofluoroalkane (HFA) MDI [90 mcg ex-actuator] or equivalent) for use on an as-needed basis for the immediate relief of asthma symptoms throughout the treatment period.
- BDP 320 mcg MDI; BDP 640 mcg MDI: Beclomethasone dipropionate (BDP) via metered dose inhaler (MDI) twice daily.
  Placebo BAI for blinding.
  Rescue medication (albuterol/salbutamol hydrofluoroalkane (HFA) MDI [90 mcg ex-actuator] or equivalent) for use on an as-needed basis for the immediate relief of asthma symptoms throughout the treatment period.
- Total: Total of all reporting groups
Arm/Group | Placebo BAI and MDI | BDP 320 mcg BAI | BDP 640 mcg BAI | BDP 320 mcg MDI | BDP 640 mcg MDI | Total
Number analyzed (Participants) | 106 | 106 | 106 | 107 | 107 | 532
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4 | 5 | 7 | 4 | 6 | 26
  Between 18 and 65 years | 94 | 86 | 92 | 93 | 92 | 457
  >=65 years | 8 | 15 | 7 | 10 | 9 | 49
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68 | 69 | 67 | 65 | 66 | 335
  Male | 38 | 37 | 39 | 42 | 41 | 197
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 6 | 3 | 5 | 2 | 2 | 18
  Black or African American | 27 | 18 | 14 | 16 | 24 | 99
  White | 73 | 85 | 87 | 89 | 81 | 415
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Standardized Baseline-adjusted Trough Morning Forced Expiratory Volume in 1 Second (FEV1) Area Under the Effect Curve From Time 0 to 12 Weeks (AUEC(0-12wk) )
Description: Trough morning FEV1 measurements were taken pre-dose and pre-rescue bronchodilator treatment for asthma. The baseline pulmonary function measurement was defined as the measurement obtained at randomization visit (Day 1). Pulmonary function measurements (including FEV1) were obtained electronically by spirometry. All pulmonary function test data were submitted to a central reading center for evaluation. The highest FEV1 value from 3 acceptable and 2 repeatable maneuvers (maximum of 5 attempts) was used.
  Baseline-adjusted FEV1 AUEC(0-12wk) were calculated using the trapezoidal rule.
  The standardized baseline-adjusted FEV1 AUEC(0-12 wk) accommodates participants who dropped out of the study. Baseline-adjusted FEV1 AUEC(0-t weeks)/t, where t =12 weeks for patients who complete the FEV1 assessment at Week 12. For participants who dropped out early, t <12 weeks (2, 4, or 8 weeks).
Time Frame: Day 1 (baseline), Weeks 2, 4, 8, 12
Population: Full analysis set- randomized patients with at least 1 dose of drug and 1 postbaseline trough am FEV1
Measure: Least Squares Mean (Standard Error); unit: Liters
Groups:
- BDP 320 mcg BAI; BDP 640 mcg BAI: Beclomethasone dipropionate (BDP) via breath-actuated inhaler (BAI) twice daily.
  Placebo MDI for blinding.
  Albuterol/salbutamol: Rescue medication (albuterol/salbutamol hydrofluoroalkane (HFA) MDI [90 mcg ex-actuator] or equivalent) for use on an as-needed basis for the immediate relief of asthma symptoms throughout the treatment period.
- BDP 320 mcg MDI; BDP 640 mcg MDI: Beclomethasone dipropionate (BDP) via metered dose inhaler (MDI) twice daily.
  Placebo BAI for blinding.
  Albuterol/salbutamol: Rescue medication (albuterol/salbutamol hydrofluoroalkane (HFA) MDI [90 mcg ex-actuator] or equivalent) for use on an as-needed basis for the immediate relief of asthma symptoms throughout the treatment period.
Arm/Group | Placebo BAI and MDI | BDP 320 mcg BAI | BDP 640 mcg BAI | BDP 320 mcg MDI | BDP 640 mcg MDI
Number analyzed (Participants) | 105 | 104 | 106 | 106 | 107
Liters | 0.056 (0.0219) | 0.09 (0.0221) | 0.101 (0.0221) | 0.041 (0.0217) | 0.096 (0.0216)
Statistical Analysis 1: Comparison: Placebo BAI and MDI vs BDP 320 mcg BAI; Test type: Superiority; p = 0.272, ANCOVA; Least Square Mean (LSM) Difference = 0.034, 95% CI 2-sided [-0.027 to 0.095]
Statistical Analysis 2: Comparison: Placebo BAI and MDI vs BDP 640 mcg BAI; Test type: Superiority; p = 0.1415, ANCOVA; LSM Difference = 0.045, 95% CI 2-sided [-0.015 to 0.106]
Statistical Analysis 3: Comparison: Placebo BAI and MDI vs BDP 320 mcg MDI; Test type: Superiority; p = 0.6356, ANCOVA; LSM Difference = -0.015, 95% CI 2-sided [-0.075 to 0.046]
Statistical Analysis 4: Comparison: Placebo BAI and MDI vs BDP 640 mcg MDI; Test type: Superiority; p = 0.1932, ANCOVA; LSM Difference = 0.04, 95% CI 2-sided [-0.02 to 0.1]

2. Secondary Outcome: Change From Baseline in Weekly Average of Daily Trough Morning Peak Expiratory Flow (PEF) Over the 12-week Treatment Period Using a Mixed Model for Repeated Measures (MMRM)
Description: A hand-held peak flow meter was provided to patients at the screening visit and used to determine the morning and evening PEF throughout the course of the study. Daily trough morning PEF assessments were taken pre-dose and pre-rescue bronchodilator over the 12-week treatment period. The patient recorded the highest value of 3 measurements obtained in the morning and evening in the patient diary.
  Baseline in trough morning PEF is defined as the average of recorded trough morning PEF assessments over the 7-day window before randomization, including the morning assessment on Day 1 before randomization.
  Weekly average PEF data was generated using 7-day windows based on analysis days (before the first dose of double-blind study treatment). PEF over the 12 week treatment period was performed using a mixed-model for repeated measures (MMRM) with effects due to baseline weekly average of daily trough morning PEF, sex, age, treatment, time, and time by treatment interaction.
Time Frame: Baseline: Days -6 to Day 1 (pre-randomization), Treatment: Day 2 to Week 12
Population: Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: Liters/minute
Groups:
- BDP 640 mcg BAI: Beclomethasone dipropionate (BDP) via breath-actuated inhaler (BAI) twice daily.
  Placebo MDI for blinding.
  Rescue medication (albuterol/salbutamol hydrofluoroalkane (HFA) MDI [90 mcg ex-actuator] or equivalent) for use on an as-needed basis for the immediate relief of asthma symptoms throughout the treatment period.
Arm/Group | Placebo BAI and MDI | BDP 320 mcg BAI | BDP 640 mcg BAI | BDP 320 mcg MDI | BDP 640 mcg MDI
Number analyzed (Participants) | 106 | 104 | 106 | 106 | 107
Liters/minute | -5.524 (2.5944) | 5.092 (2.5625) | 2.895 (2.559) | 0.480 (2.558) | 6.988 (2.5298)
Statistical Analysis 1: Comparison: Placebo BAI and MDI vs BDP 320 mcg BAI; Test type: Other — The analysis of change from baseline in weekly average of daily trough morning (pre-dose and pre-rescue bronchodilator) PEF over the 12-week treatment period was performed using a repeated measures mixed model with effects due to baseline weekly average of daily trough morning PEF, sex, age, treatment, time, and time-by-treatment interaction; p = 0.0036, Mixed Model for repeated measures; LSM Difference = 10.616, 95% CI 2-sided [3.489 to 17.744]
Statistical Analysis 2: Comparison: Placebo BAI and MDI vs BDP 640 mcg BAI; The analysis of change from baseline in weekly average of daily trough morning (pre-dose and pre-rescue bronchodilator) PEF over the 12-week treatment period was performed using a repeated measures mixed model with effects due to baseline weekly average of daily trough morning PEF, sex, age, treatment, time, and time-by-treatment interaction; Test type: Superiority; p = 0.0204, Mixed Model for repeated measures; LSM Difference = 8.419, 95% CI 2-sided [1.309 to 15.53]
Statistical Analysis 3: Comparison: Placebo BAI and MDI vs BDP 320 mcg MDI; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p = 0.0984, Mixed Model for repeated measures; LSM Difference = 6.004, 95% CI 2-sided [-1.121 to 13.129]
Statistical Analysis 4: Comparison: Placebo BAI and MDI vs BDP 640 mcg BAI; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p = 0.0006, Mixed Model for repeated measures; LSM Difference = 12.512, 95% CI 2-sided [5.435 to 19.589]

3. Secondary Outcome: Change From Baseline in Weekly Average of Daily Evening Peak Expiratory Flow (PEF) Over the 12-week Treatment Period Using a Mixed Model for Repeated Measures (MMRM)
Description: A hand-held peak flow meter was provided to patients at the screening visit and used to determine the morning and evening PEF throughout the course of the study. The patient recorded the highest value of 3 measurements obtained in the morning and evening in the patient diary.
  Baseline in evening PEF is defined as the average of recorded evening PEF assessments over the 7-day window before randomization.
  Weekly average PEF data was generated using 7-day windows based on analysis days (after the first dose of double-blind study treatment). PEF over the 12 week treatment period was performed using a mixed-model for repeated measures (MMRM) with effects due to baseline weekly average of daily evening peak PEF, sex, age, treatment, time, and time by treatment interaction.
Time Frame: Baseline: Days -7 to Day -1, Treatment: Day 1 to Week 12
Population: Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: Liters/minute
Arm/Group | Placebo BAI and MDI | BDP 320 mcg BAI | BDP 640 mcg BAI | BDP 320 mcg MDI | BDP 640 mcg MDI
Number analyzed (Participants) | 106 | 104 | 106 | 106 | 107
Liters/minute | -4.708 (2.6503) | 4.439 (2.6199) | 4.462 (2.6092) | -0.62 (2.6145) | 5.594 (2.5848)
Statistical Analysis 1: Comparison: Placebo BAI and MDI vs BDP 320 mcg BAI; Test type: Superiority; p = 0.0139, Mixed Model for repeated measures; LSM Difference = 9.147, 95% CI 2-sided [1.866 to 16.429]
Statistical Analysis 2: Comparison: Placebo BAI and MDI vs BDP 640 mcg BAI; Test type: Superiority; p = 0.0133, Mixed Model for repeated measures; LSM Difference = 9.17, 95% CI 2-sided [1.914 to 16.425]
Statistical Analysis 3: Comparison: Placebo BAI and MDI vs BDP 320 mcg MDI; Test type: Superiority; p = 0.2704, Mixed Model for repeated measures; LSM Difference = 4.088, 95% CI 2-sided [-3.191 to 11.367]
Statistical Analysis 4: Comparison: Placebo BAI and MDI vs BDP 640 mcg MDI; Test type: Superiority; p = 0.0053, Mixed Model for repeated measures; LSM Difference = 10.301, 95% CI 2-sided [3.073 to 17.53]

4. Secondary Outcome: Change From Baseline in the Weekly Average of Total Daily (24-hour) Use of Albuterol/Salbutamol Inhalation Aerosol (Number of Inhalations) Over Weeks 1-12 Using a Mixed Model for Repeated Measures (MMRM)
Description: Change from baseline in the use of rescue medication, albuterol/salbutamol, during the treatment period offers an indication of asthma control. Baseline was defined as the average of recorded daily usage of albuterol/salbutamol inhalation aerosol over the 7 days prior to the first dose of double-blind study treatment, including the morning usage at the randomization visit.
  Weekly average rescue medication data was generated using 7-day windows based on analysis days (after the first dose of double-blind study treatment). Weekly average over the 12 week treatment period was performed using a mixed-model for repeated measures (MMRM) with effects due to baseline value, sex, age, time, treatment, and time-by-treatment interaction.
Time Frame: Baseline: Days -6 to Day 1 (pre-randomization), Treatment: Day 1 to Week 12
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: number of inhalations
Arm/Group | Placebo BAI and MDI | BDP 320 mcg BAI | BDP 640 mcg BAI | BDP 320 mcg MDI | BDP 640 mcg MDI
Number analyzed (Participants) | 101 | 96 | 99 | 97 | 101
number of inhalations | 0.478 (0.1232) | -0.226 (0.1235) | -0.213 (0.1221) | -0.173 (0.1246) | -0.323 (0.1206)
Statistical Analysis 1: Comparison: Placebo BAI and MDI vs BDP 320 mcg BAI; Test type: Superiority; p < 0.0001, Mixed Model for repeated measures; LSM Difference = -0.703, 95% CI 2-sided [-1.044 to -0.363]
Statistical Analysis 2: Comparison: Placebo BAI and MDI vs BDP 640 mcg BAI; Test type: Superiority; p < 0.0001, Mixed Model for repeated measures; LSM Difference = -0.691, 95% CI 2-sided [-1.029 to -0.352]
Statistical Analysis 3: Comparison: Placebo BAI and MDI vs BDP 320 mcg MDI; Test type: Superiority; p = 0.0002, Mixed Model for repeated measures; LSM Difference = -0.651, 95% CI 2-sided [-0.994 to -0.309]
Statistical Analysis 4: Comparison: Placebo BAI and MDI vs BDP 640 mcg MDI; Test type: Superiority; p < 0.0001, Mixed Model for repeated measures; LSM difference = -0.801, 95% CI 2-sided [-1.138 to -0.464]

5. Secondary Outcome: Change From Baseline in the Weekly Average of the Total Daily Asthma Symptom Score Over Weeks 1-12 Using a Mixed Model for Repeated Measures (MMRM)
Description: Asthma symptom scores are recorded in the patient's diary each morning and each evening before determining PEF and before administration of study or rescue medications. The Daytime Symptom Score (determined in the evening) has a range from 0=No symptoms during the day to 5=Symptoms so severe that I could not go to work or perform normal daily activities. The Nighttime Symptom Score (determined in the morning) has a range from 0=No symptoms during the night to 4=Symptoms so severe that I did not sleep at all. The total daily asthma symptom score is the average of the daytime and the nighttime scores (full scale is 0 - 4.5). The total daily asthma symptom score is missing if either the daytime or nighttime score is missing. Baseline was the average of recorded daily asthma symptom scores over 7 days prior to the first dose of study treatment. The weekly average was the sum of total daily asthma symptom scores over the 7 days divided by the number of non-missing assessments.
Time Frame: Days -6 to Day 1 (pre-randomization), Treatment: Day 1 to Week 12
Population: Full analysis set. Analysis used a MMRM with effects due to baseline score, sex, age, time, treatment, and time-by-treatment interaction.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo BAI and MDI | BDP 320 mcg BAI | BDP 640 mcg BAI | BDP 320 mcg MDI | BDP 640 mcg MDI
Number analyzed (Participants) | 106 | 104 | 106 | 106 | 107
units on a scale | -0.058 (0.0425) | -0.207 (0.0417) | -0.159 (0.0415) | -0.247 (0.0417) | -0.274 (0.0411)
Statistical Analysis 1: Comparison: Placebo BAI and MDI vs BDP 320 mcg BAI; Test type: Superiority; p = 0.0119, Mixed Models Analysis; Mean Difference (Final Values) = -0.149, 95% CI 2-sided [-0.265 to -0.033]
Statistical Analysis 2: Comparison: Placebo BAI and MDI vs BDP 640 mcg BAI; Test type: Superiority; p = 0.0854, Mixed Models Analysis; Mean Difference (Final Values) = -0.102, 95% CI 2-sided [-0.217 to 0.014]
Statistical Analysis 3: Comparison: Placebo BAI and MDI vs BDP 320 mcg MDI; Test type: Superiority; p = 0.0016, Mixed Models Analysis; Mean Difference (Final Values) = -0.189, 95% CI 2-sided [-0.306 to -0.072]
Statistical Analysis 4: Comparison: Placebo BAI and MDI vs BDP 640 mcg MDI; Test type: Superiority; p = 0.0003, Mixed Models Analysis; Mean Difference (Final Values) = -0.216, 95% CI 2-sided [-0.332 to -0.101]

6. Secondary Outcome: Kaplan-Meier Estimates for Time to Withdrawal From Study Treatment Due to Meeting Stopping Criteria for Worsening Asthma
Description: Time to withdrawal due to meeting stopping criteria is defined as number of days elapsed from the date of the first dose of double-blind study treatment to the date of withdrawal due to meeting stopping criteria. Stopping criteria are:
  * FEV1 as measured at the study center is below the FEV1 stability limit value calculated at RV.
  * Based upon review of patient diary data, the patient has experienced any of the following during any 7-day period:
  * 4+ days in which the highest (of 3 efforts) am PEF fall below the PEF stability limit calculated when randomized. The patient meets with the investigator who determines whether the FEV1 is consistent with worsening asthma;
  * 3+ days in which 12+ inhalations/day of rescue medication were used
  * 2+ days in which the patient experienced a nighttime asthma symptom score of more than 2
  * Clinical asthma exacerbation requiring (for example) the use of systemic corticosteroids, or the emergency room or hospitalization.
Time Frame: Day 1 - Week 12
Population: Full analysis set; unable to calculate as few patients met stopping criteria
Measure: Median (95% Confidence Interval); unit: days
Groups:
- Placebo BAI or MDI: Placebo breath-actuated inhaler (BAI), twice daily. Plus placebo metered dose inhaler (MDI), twice daily.
  Rescue medication (albuterol/salbutamol hydrofluoroalkane (HFA) MDI [90 mcg ex-actuator] or equivalent) for use on an as-needed basis for the immediate relief of asthma symptoms throughout the treatment period.
Arm/Group | Placebo BAI or MDI | BDP 320 mcg BAI | BDP 640 mcg BAI | BDP 320 mcg MDI | BDP 640 mcg MDI
Number analyzed (Participants) | 106 | 104 | 106 | 106 | 107
days | NA [NA to NA] — The median and 95% CI of the median is not applicable if the proportion of participants withdrawn is less than 0.5. | NA [NA to NA] — The median and 95% CI of the median is not applicable if the proportion of participants withdrawn is less than 0.5. | NA [NA to NA] — The median and 95% CI of the median is not applicable if the proportion of participants withdrawn is less than 0.5. | NA [NA to NA] — The median and 95% CI of the median is not applicable if the proportion of participants withdrawn is less than 0.5. | NA [NA to NA] — The median and 95% CI of the median is not applicable if the proportion of participants withdrawn is less than 0.5.

7. Secondary Outcome: Number of Participants Withdrawn From Study Due to Meeting Stopping Criteria for Worsening Asthma During the 12-Week Treatment Period
Description: A count of participants who were withdrawn from the study due to meeting stopping criteria. Alert criteria for individual patients with worsening asthma were designed to ensure patient safety. The investigator determined whether the patient's overall clinical picture is consistent with worsening asthma and if the patient should be withdrawn from study drug treatment (but not the study) and be placed on appropriate asthma therapy in the interest of patient safety.
  An example of alert criteria is:
  * FEV1 as measured at the study center is below the FEV1 stability limit value calculated at randomization visit (Day 1).
  * Other criteria as defined in the protocol.
Time Frame: Treatment period: Day 1 up to Week 12
Population: Full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo BAI or MDI | BDP 320 mcg BAI | BDP 640 mcg BAI | BDP 320 mcg MDI | BDP 640 mcg MDI
Number analyzed (Participants) | 106 | 104 | 106 | 106 | 107
Participants | 15 | 3 | 3 | 5 | 1

ADVERSE EVENTS:
Time Frame: - Run-In Period: Days -21 to Day 1 - Double-blind Treatment Period: Day 1 to Week 12
Groups:
- BAI 640 mcg/Day: Beclomethasone dipropionate (BDP) via breath-actuated inhaler (BAI) twice daily.
  Placebo MDI for blinding. Rescue medication (albuterol/salbutamol hydrofluoroalkane (HFA) MDI [90 mcg ex-actuator] or equivalent) for use on an as-needed basis for the immediate relief of asthma symptoms.
- MDI 320 mcg/Day; MDI 640 mcg/Day: Beclomethasone dipropionate (BDP) via metered dose inhaler (MDI) twice daily. Placebo BAI for blinding. Rescue medication (albuterol/salbutamol hydrofluoroalkane (HFA) MDI [90 mcg ex-actuator] or equivalent) for use on an as-needed basis for the immediate relief of asthma symptoms.
- Run-in Period Experience for Randomized Participants: Experience of randomized participants during the Run-In Period when they were administered standard ICS (fluticasone propionate) as well as single-blind placebo BAI and single-blind placebo MDI devices for twice-daily use.
Arm/Group | BDP 320 mcg BAI | BAI 640 mcg/Day | MDI 320 mcg/Day | MDI 640 mcg/Day | Placebo BAI and MDI | Run-in Period Experience for Randomized Participants
All-Cause Mortality (participants affected / at risk) | 0/106 | 0/106 | 0/107 | 0/107 | 0/106 | 0/532
Serious Adverse Events (participants affected / at risk) | 1/106 | 1/106 | 1/107 | 2/107 | 0/106 | 1/532
Other Adverse Events (participants affected / at risk) | 9/106 | 11/106 | 9/107 | 12/107 | 2/106 | 8/532
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BDP 320 mcg BAI (N=106) | BAI 640 mcg/Day (N=106) | MDI 320 mcg/Day (N=107) | MDI 640 mcg/Day (N=107) | Placebo BAI and MDI (N=106) | Run-in Period Experience for Randomized Participants (N=532)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diverticular perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastric disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngeal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BDP 320 mcg BAI (N=106) | BAI 640 mcg/Day (N=106) | MDI 320 mcg/Day (N=107) | MDI 640 mcg/Day (N=107) | Placebo BAI and MDI (N=106) | Run-in Period Experience for Randomized Participants (N=532)
Oral candidiasis (Infections and infestations) | 5 (7) | 10 (12) | 3 (3) | 9 (11) | 0 (0) | 7 (7)
Upper respiratory tract infection (Infections and infestations) | 4 (4) | 1 (1) | 7 (7) | 4 (4) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.